CLINICAL TRIAL: NCT04178200
Title: Evaluation of Duration of Anesthesia and Patient Satisfaction After Retrobulbar Block Applied in Cataract Surgery
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Develi Devlet Hastanesi (Other Government)
Responsible Party: Principal Investigator, Gamze ALBAYRAK, Clinical Specialist Doctor, Develi Devlet Hastanesi
Other Study IDs: 2019/776
Record Dates: First submitted 2019-11-20; First posted 2019-11-26 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Cataract Surgery; Patient Satisfaction; Akinesia; Anesthesia, Local; Anesthesia; Adverse Effect; Anesthesia Recovery Period
Keywords: Cataract; Retrobulbar Block; Ocular and eyelid; Akinesia; Anesthesia Recovery Period; Patient Satisfaction; Pain Score
MeSH Terms: conditions — Patient Satisfaction; Cataract | interventions — Lidocaine; Bupivacaine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- 1.5 ml Dose: For retrobulbar anesthesia, 1.5 ml of local anesthetic solution (2% lidocaine, 5% bupivacaine) will be administered to the patients.
  Interventions: Drug: Lidocaine 2% Injectable Solution 0.75 ml; Drug: Bupivacaine Hcl 0.5% Inj 0.75 ml
- 3 ml Dose: For retrobulbar anesthesia, 3 ml of local anesthetic solution (2% lidocaine, 5% bupivacaine) will be administered to the patients.
  Interventions: Drug: Lidocaine 2% Injectable Solution 1.5 ml; Drug: Bupivacaine Hcl 0.5% Inj 1.5 ml

INTERVENTIONS:
Drug: Lidocaine 2% Injectable Solution 0.75 ml — 0.75 ml of Lidocaine will be added to the anesthetic solution.
  Other Names: Lidocaine
  Groups: 1.5 ml Dose
Drug: Bupivacaine Hcl 0.5% Inj 0.75 ml — 0.75 ml of Bupivacaine will be added to the anesthetic solution.
  Other Names: Bupivacaine
  Groups: 1.5 ml Dose
Drug: Lidocaine 2% Injectable Solution 1.5 ml — 1.5 ml of Lidocaine will be added to the anesthetic solution.
  Other Names: Lidocaine
  Groups: 3 ml Dose
Drug: Bupivacaine Hcl 0.5% Inj 1.5 ml — 1.5 ml of Bupivacaine will be added to the anesthetic solution.
  Other Names: Bupivacaine
  Groups: 3 ml Dose

SUMMARY:
It is aimed to determine patient satisfaction (pain assessment during and after the operation) and the initial and total anesthesia durations of eye lid and globe anesthesia after administration of local anesthetic solution only in standard applied volumes (1.5-3 ml). No agents will be added to the local anesthetic agents used in the conventional retrobulbar block in patients who will undergo cataract surgery,

DETAILED DESCRIPTION:
In this study, 80 patients with American Society of Anesthesiologists (ASA) I-II-III who accepted retrobulbar anesthesia before cataract surgery and who were over 18 years of age and under 90 years of age were included in the study. Not accepting local anesthesia, being under 18 years of age, having problems in communication, having eyelid or eye anomaly, having Parkinson's disease, myopia with axial length ≥ 26 mm, hypersensitivity to local anesthetics or other drugs, and bleeding or other drug-induced clotting problem were determined as exclusion criteria for the investigator's study.

Written informed consent will be obtained from patients eligible for the study according to the above criteria. While obtaining informed consent, it will also be verbally stated that this study does not include any risks other than the risks of standard cataract surgery and retrobulbar block.

Patients taken to the operating room before the operation will be monitored and baseline blood pressure, pulse and peripheral capillary oxygen saturation (SpO2) values will be recorded. 2lt / min oxygen will be administered to patients with a nasal cannula. The normal ocular and valve movements of the patient will be checked and recorded before the procedure. Patients will receive a 20 gauge intravenous (IV) cannula. Before the retrobulbar block is applied, topical anesthesia is provided with 0.5% proparacaine drops and field cleaning with povidone iodine will be performed. The patient will be instructed to look at the finger held by the assistant personnel to bring the eyeball to the neutral position and the local anesthetic mixture will be slowly injected into the retrobulbar area with a 25 gauge ophthalmic needle. For retrobulbar anesthesia, 1.5-3 ml of local anesthetic solution (2% lidocaine, 5% bupivacaine) will be administered to the patients. The maximum treatment duration is 1 day and single dose. Gently massage the eye to disperse the local anesthetic solution and reduce bleeding. After block 1, 3, 5 and 10 minutes ocular movements and valve movements will be evaluated. To do this, patients will be told to look up, down, right and left and be asked to squeeze and open their eyelids. Ocular movements will be scored for each direction separately if normal, 2 if slightly restricted, and 0 if there is no movement (total score 0-8) [1]. In the evaluation of eye lid movements, complete immobility will be scored as 0, partial movement as 1 and normal movement as 2 [2]. The patient's blood pressure, pulse and SpO2 values will be recorded at 5 min intervals throughout the operation. During the operation, the pain of the patients will be assessed by a 3-point scale (0: no pain; 1: uncomfortable; 3: pain). Postoperative ocular and eye lid akinesia scores of the patients will be recorded at 30-minute intervals. Ocular and eye lid akinesia times will be recorded. Any side effects that occur during and after the procedure will be recorded. One day later, patients' responses will be recorded by asking for the first time and the number of times they need analgesics.

ELIGIBILITY:
Inclusion Criteria:

1. To accept retrobulbar anesthesia before cataract surgery
2. To be over 18 and under 90
3. Being ASA I-II-III

Exclusion Criteria:

1. Not to accept local anesthesia
2. To be under 18 years
3. Having problems in communication
4. To have lid or eye anomaly
5. Being Parkinson's
6. Being myopia with axial length ≥ 26 mm
7. Hypersensitivity to local anesthetics or other drugs
8. Having bleeding or other drug related clotting problems

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 80 people will be included in the study. All adult patients of ASA (American Society of Anesthesiologists) I-II-III who accept retrobulbar anesthesia before cataract surgery will be included in the study.
  The study will not include a vulnerable population, such as people with disabilities, children, pregnant women, puerperants and nursing women, people in intensive care and unconscious, and those who cannot give consent in person or vulnerable subjects.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2019-12-16 (Estimated); Primary Completion 2020-04-24 (Estimated); Study Completion 2020-04-24 (Estimated)

PRIMARY OUTCOMES:
Patient Pain Score | Immediately after the surgery
  patient pain assessed by with pain score of 3 points-scale (0 No pain,1 Not comfortable, 2 Have pain )
The scores of ocular and eyelid movements | at 1 minutes after the block
  Ocular movements will be scored separately for each direction, 2 if normal, 1 if slightly restricted and 0 if no movement. Complete inactivity will be scored as 0, partial movement as 1, and normal movement as 2 in the evaluation of eyelid movements.
The scores of ocular and eyelid movements | at 3 minutes after the block
  Ocular movements will be scored separately for each direction, 2 if normal, 1 if slightly restricted and 0 if no movement. Complete inactivity will be scored as 0, partial movement as 1, and normal movement as 2 in the evaluation of eyelid movements.
The scores of ocular and eyelid movements | at 5 minutes after the block
  Ocular movements will be scored separately for each direction, 2 if normal, 1 if slightly restricted and 0 if no movement. Complete inactivity will be scored as 0, partial movement as 1, and normal movement as 2 in the evaluation of eyelid movements.
The scores of ocular and eyelid movements | at 10 minutes after the block
  Ocular movements will be scored separately for each direction, 2 if normal, 1 if slightly restricted and 0 if no movement. Complete inactivity will be scored as 0, partial movement as 1, and normal movement as 2 in the evaluation of eyelid movements.
The postoperative scores of ocular and eyelid movements | at 30 minutes after the operation
  Ocular movements will be scored separately for each direction, 2 if normal, 1 if slightly restricted and 0 if no movement. Complete inactivity will be scored as 0, partial movement as 1, and normal movement as 2 in the evaluation of eyelid movements.
The postoperative scores of ocular and eyelid movements | at 60 minutes after the operation
  Ocular movements will be scored separately for each direction, 2 if normal, 1 if slightly restricted and 0 if no movement. Complete inactivity will be scored as 0, partial movement as 1, and normal movement as 2 in the evaluation of eyelid movements.
The postoperative scores of ocular and eyelid movements | at 90 minutes after the operation
  Ocular movements will be scored separately for each direction, 2 if normal, 1 if slightly restricted and 0 if no movement. Complete inactivity will be scored as 0, partial movement as 1, and normal movement as 2 in the evaluation of eyelid movements.
The postoperative scores of ocular and eyelid movements | at 120 minutes after the operation
  Ocular movements will be scored separately for each direction, 2 if normal, 1 if slightly restricted and 0 if no movement. Complete inactivity will be scored as 0, partial movement as 1, and normal movement as 2 in the evaluation of eyelid movements.
The postoperative scores of ocular and eyelid movements | at 150 minutes after the operation
  Ocular movements will be scored separately for each direction, 2 if normal, 1 if slightly restricted and 0 if no movement. Complete inactivity will be scored as 0, partial movement as 1, and normal movement as 2 in the evaluation of eyelid movements.
The postoperative scores of ocular and eyelid movements | at 180 minutes after the operation
  Ocular movements will be scored separately for each direction, 2 if normal, 1 if slightly restricted and 0 if no movement. Complete inactivity will be scored as 0, partial movement as 1, and normal movement as 2 in the evaluation of eyelid movements.
The postoperative scores of ocular and eyelid movements | at 210 minutes after the operation
  Ocular movements will be scored separately for each direction, 2 if normal, 1 if slightly restricted and 0 if no movement. Complete inactivity will be scored as 0, partial movement as 1, and normal movement as 2 in the evaluation of eyelid movements.
The scores of ocular and eyelid movements | at 240 minutes after the operation
  Ocular movements will be scored separately for each direction, 2 if normal, 1 if slightly restricted and 0 if no movement. Complete inactivity will be scored as 0, partial movement as 1, and normal movement as 2 in the evaluation of eyelid movements.

SECONDARY OUTCOMES:
The need for analgesic and how many times it needs | One day after the surgery
  The patients will be asked whether they need analgesia (yes or no), if they need analgesia, they will be asked what time and how many times they take analgesic agents.
side effects questionnaire | One day after the surgery
  Ophthalmic side effects (Globe perforation, Pain at the injection site, Pressure sensation behind the eye, Subconjunctival hemorrhage, Retrobulbar hemorrhage, hematoma, ecchymosis, diplopia, ptosis) and other side effects (Nausea and vomiting, arrhythmia, Convulsion, Allergy, Weakness)

CONTACTS AND LOCATIONS:
Overall Officials: Gamze ALBAYRAK, MD, Principal Investigator — Develi Devlet Hastanesi
Locations (1):
- Develi Hatice Muammer Kocatürk Devlet Hastanesi, Develi, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barr J, Kirkpatrick N, Dick A, Leonard L, Hawksworth G, Noble DW. Effects of adrenaline and hyaluronidase on plasma concentrations of lignocaine and bupivacaine after peribulbar anaesthesia. Br J Anaesth. 1995 Dec;75(6):692-7. doi: 10.1093/bja/75.6.692. PMID 8672315
- [Background] Sarvela PJ. Comparison of regional ophthalmic anesthesia produced by pH-adjusted 0.75% and 0.5% bupivacaine and 1% and 1.5% etidocaine, all with hyaluronidase. Anesth Analg. 1993 Jul;77(1):131-4. doi: 10.1213/00000539-199307000-00026. PMID 8317720